CLINICAL TRIAL: NCT05607758
Title: Digital Stress Management Intervention for Health Care Providers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Elin Børøsund, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22/21663
Record Dates: First submitted 2022-11-02; First posted 2022-11-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Health Care Providers; Stress; Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App for Stress management (Experimental): Participants will:
  * Participate in a physical introduction to the app-based stress management program
  * Get access to the app-based program, and a new module every third day (total 10 modules). The app consists of stress management education, cognitive behavioral interventions and relaxation training exercises.
  * Receive two phone follow-up calls from study personnel (about 3 and 6 weeks after the physical introduction)
  Interventions: Behavioral: StressProffen©™

INTERVENTIONS:
Behavioral: StressProffen©™ — An app-based program for stress management consisting of 10 modules that teaches stress management, cognitive behavioral coping skills and relaxation training.
  Other Names: Stress Management

SUMMARY:
The purpose with this study is to test if the app-based stress management program StressProffen, can be of interest and support for stress management among health care providers.

DETAILED DESCRIPTION:
For health care providers, work-related stress can be a major challenge that can lead to frustration, lower motivation, reduced quality of life and burnout, and the last year's COVID-19 pandemic particularly emphasized the challenges in the stressful everyday life faced by health care providers.

There are, however, interventions that can be of support, both for the prevention of stress and for coping with stress in challenging situations, and in recent years there has also been an increased focus on stress in working life in this setting. Several studies have also recently been carried out which aim to deliver such interventions via applications (apps) to promote employees' physical and mental health, as well as their ability to cope with stress. However, there is a need for more research in the field, especially with a focus that content in such apps should be based on evidence-based theory, and that interviews and a similar qualitative approach should be included in studies to gain increased insight into the need for and usefulness of digital tools among health care providers.

This study will therefore test the effect of an app-based program for stress management, StressProffen, among health care providers, in a single arm study. The app contains 10 modules distributed over four weeks, focusing on education of different techniques for reduction of stress and stress reduction exercises.

StressProffen was initially developed and tested for stress management in patients with cancer, with good results. Among other things, a randomized controlled trial showed a statistically significant reduction in perceived stress, anxiety, depression and self-regulation fatigue, as well as increased health-related quality of life, for participants in the intervention group compared to the control group. The aim of this study is to test whether StressProffen can be of interest and support for stress management among health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Health care providers (included but not restricted to, registered nurses, physicians, physiotherapists, occupational therapists, dietitians, social workers, health workers).
* Working with patient treatment or follow up at Oslo University Hospital
* Having their own smart phone or tablet
* Being able to write/read/speak Norwegian

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The Perceived Stress Scale (PSS-14) | Change from baseline to f-up month 3
  14 item scale measuring perceived stress. Scale range: 0-56. Higher scores indicate higher perceived stress.
The Perceived Stress Scale (PSS-14) | Change from baseline to f-up month 6
  14 item scale measuring perceived stress. Scale range: 0-56. Higher scores indicate higher perceived stress.

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) | Change from baseline to f-up month 3
  14 item scale measuring anxiety and depression. The Scale has a total score with a scale range of 0 to 42 and an anxiety (HADS-A) and a depression (HADS-D) subscale, both with scale range of 0 to 21.
  Sub scale scores: 0-7= Normal, 8-10= Borderline abnormal (borderline case), 11-21= abnormal (case).
The Hospital Anxiety and Depression Scale (HADS) | Change from baseline to f-up month 6
  14 item scale measuring anxiety and depression. The Scale has a total score with a scale range of 0 to 42 and an anxiety (HADS-A) and a depression (HADS-D) subscale, both with scale range of 0 to 21.
  Sub scale scores: 0-7= Normal, 8-10= Borderline abnormal (borderline case), 11-21= abnormal (case).
SF-36 Item Short Form Health Survey (RAND-36 version) | Change from baseline to f-up month 3
  36 item scale measuring health related quality of life (HRQoL). The scale has 8 subscales and 1 single item score. Scale and single item range: 0 to 100. Higher scores indicate higher HRQoL.
SF-36 Item Short Form Health Survey (RAND-36 version) | Change from baseline to f-up month 6
  36 item scale measuring health related quality of life (HRQoL). The scale has 8 subscales and 1 single item score. Scale and single item range: 0 to 100. Higher scores indicate higher HRQoL.
The Self-Regulatory Fatigue-18 (SRF-18) | Change from baseline to f-up month 3
  18 item scale measuring self-regulation. Scale range: 18 to 90. A higher score indicates higher self-regulatory fatigue
The Self-Regulatory Fatigue-18 (SRF-18) | Change from baseline to f-up month 6
  18 item scale measuring self-regulation. Scale range: 18 to 90. A higher score indicates higher self-regulatory fatigue

OTHER OUTCOMES:
Intervention commentary | 3 months
  A six item brief measure of participant's intervention reactions. The first 3 items gauged participants' program perception on a scale from 1 to 5, with 5 indicating better perception. The next 3 items were open ended questions: * What did you like best? * What did you like the least? * Suggestions for improvement?
Sleep | Change from baseline to f-up month 3
  Four questions related to number of hours of sleep per 24 hours, how much sleep participants need to feel rested, experienced quality of sleep an impact of shift-work on sleep
Sleep | Change from baseline to f-up month 6
  Four questions related to number of hours of sleep per 24 hours, how much sleep participants need to feel rested, experienced quality of sleep an impact of shift-work on sleep

CONTACTS AND LOCATIONS:
Overall Officials: Lise Solberg Nes, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No